CLINICAL TRIAL: NCT03084172
Title: Systemic Redesign and Demonstration for Early Detection, Evaluation and Management of Chronic Kidney Disease in Shanghai
Acronym: SCREENING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Shanghai Municipal Commission of Health and Family Planning (Other); Shanghai Municipal Center for Disease Control and Prevention (Other); Huashan Hospital (Other); Shanghai Minhang district Municipal Center for Disease Control and Prevention (Unknown); Shanghai Jing'an district Municipal Center for Disease Control and Prevention (Unknown); Fudan University (Other); Minhang District Central Hospital of Shanghai (Unknown); Jing'an District Central Hospital of Shanghai (Unknown); Jing'an District Zhabei Central Hospital of Shanghai (Unknown); Jing'an District Shibei Hospital of Shanghai (Unknown); Linfen Community Health Services Center of Shanghai (Unknown); Pengpu Community Health Services Center of Shanghai (Unknown); Pengpu zhen Community Health Services Center of Shanghai (Unknown); Da'ning Community Health Services Center of Shanghai (Unknown); Gonghexin Community Health Service Center of Shanghai (Unknown); Zhijiangxi Road Community Health Service Center of Shanghai (Unknown); Tianmuxi Road Community Health Service Center of Shanghai (Unknown); Beizhan Community Health Service Center of Shanghai (Unknown); Baoshan Community Health Services Center of Shanghai (Unknown); West Nanjing road Community Health Services Center of Shanghai (Unknown); Second Shimen Road Community Health Service Center of Shanghai (Unknown); Jiangning Road Community Health Service Center of Shanghai (Unknown); Caojiadu Community Health Service Center of Shanghai (Unknown); Jing'an Temple Community Health Service Center of Shanghai (Unknown); Xinzhuang Community Health Service Center of Shanghai (Unknown); Longbai Community Health Service Center of Shanghai (Unknown); Gumei Community Health Service Center of Shanghai (Unknown); Xinhong Community Health Service Center of Shanghai (Unknown); Huacao Community Health Service Center of Shanghai (Unknown); Hongqiao Community Health Service Center of Shanghai (Unknown); Qibao Community Health Service Center of Shanghai (Unknown); Meilong Community Health Service Center of Shanghai (Unknown); Jiangchuan Community Health Service Center of Shanghai (Unknown); Zhuanqiao Community Health Service Center of Shanghai (Unknown); Maqiao Community Health Service Center of Shanghai (Unknown); Wujing Community Health Service Center of Shanghai (Unknown); Pujiang Community Health Service Center of Shanghai (Unknown)
Responsible Party: Principal Investigator, Changlin Mei, Professor, Director of kidney Institute of the people's Liberation Army, Shanghai Changzheng Hospital
Other Study IDs: CZKIPLA-CKD-001
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic kidney disease patients group: These patients were screened from 2000000 of the population. The investigator will compare the prevalence rate, awareness rate and treatment rate before and after the completion of the system. The degree of decreased glomerular filtration rate is also an important evaluation index.

SUMMARY:
Based on clinical evidence based medicine and organizational management model, investigators redesign the prevention and treatment of chronic kidney disease of public health system in Shanghai China. The investigators hope to find early chronic kidney disease, prevention and clinical intervention of orderly combination. The advantages of this system were confirmed by comparing the prevalence rate, awareness rate and treatment rate before and after the completion of the system.

DETAILED DESCRIPTION:
The whole study mainly includes the following parts:

1. Establishment of a database of patients with kidney disease, and training data entry specialist in every center.
2. Conduct propaganda of kidney disease knowledge, training professional doctors in center hospital and community hospital.
3. Search for high-risk patients, and screening for patients with kidney disease from community residents in community hospital.
4. Establishment of a standardized and orderly patient referral process from community hospital to center hospital or three level of first-class hospital.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Signed informed consent

Exclusion Criteria:

* Refused to accept the blood and urine test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The residents in Jing'an District and Minhang District, which medical services are provided by those collaborative Community Health Service Center.
Sampling Method: Non-Probability Sample
Enrollment: 2000000 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
prevalence rate of chronic kidney disease | baseline and 12 months, an average of 3 years
  Change in prevalence rate of chronic kidney disease in shanghai from baseline to 3 years.
awareness rate of chronic kidney disease | baseline and 12 months, an average of 3 years
  Change in awareness rate of chronic kidney disease in shanghai from baseline to 3 years.
treatment rate of chronic kidney disease | baseline and 12 months, an average of 3 years
  Change in using standardized and orderly patient referral process from community hospital to center hospital or three level of first-class hospital. in shanghai from baseline to 3 years.
The degree of decreased glomerular filtration rate in chronic kidney patients | through study completion, an average of 3 years
  The degree of decreased glomerular filtration rate in chronic kidney patients, compared with healthy people and reported level in the literatures

CONTACTS AND LOCATIONS:
Overall Officials: Changlin Mei, Master, Principal Investigator — Shanghai Changzheng Hospital
Locations (34):
- China (34):
  - Changzheng Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Jiangning Road Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Jing'an District Central Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Jing'an Temple Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Second Shimen Road Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - West Nanjing road Community Health Services Center of Shanghai, Shanghai, Shanghai Municipality
  - Caojiadu Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Jing'an District Zhabei Central Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Tianmuxi Road Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Zhijiangxi Road Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Baoshan Community Health Services Center of Shanghai, Shanghai, Shanghai Municipality
  - Beizhan Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Da'ning Community Health Services Center of Shanghai, Shanghai, Shanghai Municipality
  - Gonghexin Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Pengpu zhen Community Health Services Center of Shanghai, Shanghai, Shanghai Municipality
  - Jiangchuan Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - The Fifth People's Hospital of Shanghai, Fudan University, Shanghai, Shanghai Municipality
  - Wujing Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Linfen Community Health Services Center of Shanghai, Shanghai, Shanghai Municipality
  - Pengpu Community Health Services Center of Shanghai, Shanghai, Shanghai Municipality
  - Jing'an District Shibei Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Minhang District Central Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Xinhong Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Xinzhuang Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Qibao Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Gumei Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Hongqiao Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Meilong Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Longbai Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Huacao Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Zhuanqiao Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Maqiao Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality
  - Pujiang Community Health Service Center of Shanghai, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No